CLINICAL TRIAL: NCT05075928
Title: Description of a Cohort of Covid-19 Patients With a Circulating Anticoagulant
Acronym: LA-COVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7861
Record Dates: First submitted 2021-10-06; First posted 2021-10-13 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-10

CONDITIONS: SARS-COV-2
Keywords: SARS-COV-2; Covid-19; Antiphospholipid syndrome (APS); autoimmune disease; antiphospholipid antibodies (aPL); thrombosis
MeSH Terms: conditions — COVID-19; Antiphospholipid Syndrome; Autoimmune Diseases; Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
SARS-COV-2 infection is responsible for a potentially severe primarily respiratory infection called COVID19. A large proportion of patients, in particular in severe forms, present with thrombotic manifestations (DVT, EP, stroke, thrombosis of dialysis circuits, etc.). A significant proportion is also a carrier of circulating anticoagulant (ACC or LA), making it possible to suggest a diagnosis of APS. This type of autoantibody results in a spontaneous prolongation of the TCA uncorrected by a control serum therefore is quickly diagnosed using standard hemostasis The objective of this study is to describe the diagnosis of thrombotic complications in COVID19 patients presenting a positive lupus anticoagulant type test (LA) or aPL and the associated clinical and biological elements that may have favored thrombosis.

ELIGIBILITY:
Inclusion criteria:

* Adult patient (≥18 years old)
* Patient taken care of in the SMO pole or the NHC surgical resuscitation service or hospitalized or consultant to the HUS between 01/03/2020 and 31/05/2020
* Patient infected with Covid-19, with a documented infection, having presented a documented thrombosis (arterial or venous), with an LA or aPL in the thrombosis assessment
* or Patient infected with Covid-19, with a documented infection, without documented thrombosis (arterial or venous), with in the standard work-up an increase in TCA revealing the presence of LA
* Subject having given his agreement for the reuse of his data for the purposes of this research

Exclusion criteria:

* Subject having expressed opposition to participating in the study
* Subject under guardianship or guardianship
* Subject under safeguard of justice

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major patient infected with Covid-19, with a documented infection, having presented a documented thrombosis (arterial or venous), with an LA or aPL in the thrombosis assessment
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Retrospective study of thrombotic complications in a cohort of COVID patients with a circulating anticoagulant | Files analysed retrospectively from March 01, 2020 to May 31, 2019 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Sophie Korganow, MD, PhD, Principal Investigator — Service de Médecine Interne et d'Immunologie Clinique - Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de Médecine Interne et d'Immunologie Clinique - Hôpitaux Universitaires de Strasbourg, Strasbourg, France